CLINICAL TRIAL: NCT06047886
Title: Feasibility Study of CD34 Selection for GVHD Prophylaxis Using the Automated CliniMACS
Brief Title: UAB 2419-CD34 Selection Using the Automated CliniMACS Prodigy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Antonio Di Stasi, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE29384
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: AML; ALL; Lymphoid Malignancies; Myelodysplastic Syndromes; CML; Primary Myelofibrosis
Keywords: hematologic malignancies; graft failure
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility study of CD34 selection for graft versus host disease (GVHD) Prophylaxis using the automated CliniMACS Prodigy Device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment population (Experimental): Patients status post allogeneic hematopoietic stem cell transplantation for a neoplastic hematologic disorder with the need of a CD34 selected stem cell boost for graft failure or low graft function will receive a CD34 selected hematopoietic stem cell infusion with or without preceding conditioning.
  Fludarabine 25 mg/mq day 1 - 5 + 2 Gray Total body irradiation depending on clinician's discretion (with the addition of cyclophosphamide 14.5 mg/kg for two doses for haploidentical or matched unrelated donor with at least one major HLA mismatch). Recommendation to use a conditioning regimen include complete loss of donor chimerism, trilineage cytopenias.
  Interventions: Drug: Infusion of CD34 selected hematopoietic stem cells

INTERVENTIONS:
Drug: Infusion of CD34 selected hematopoietic stem cells — CD34 stem cell isolation and infusion to reduce alloreactive complication of stem cell infusion

SUMMARY:
Patients with graft failure or delayed engraftment may benefit from a hematopoietic stem cell boost or an additional hematopoietic stem cell transplantation procedure. In such settings standard immune suppression strategies are avoided due to their myelosuppressive nature. Therefore those patients are at increased risk of graft versus host disease, and the infusion of a CD34 selected graft would reduce such a risk. The infusion of CD34 selected graft using CliniMACS plus is currently FDA FDA-approved indication for acute myeloid leukemia. However, the use of the Prodigy would streamline the processing, in terms of hands-off procedure, allowing to provision of this product to the patients without strains on the cell therapy lab team. This procedure has been demonstrated safe and effective in several single-center studies and is currently in advanced phase investigation in several studies for malignant and non-malignant conditions.

DETAILED DESCRIPTION:
Patients eligible to be treated on this status are status post allogeneic hematopoietic stem cell transplantation for a neoplastic hematologic disorder with the need of a CD34 selected stem cell boost for graft failure or low graft function (e.g. marrow cellularity reduced per age and/or dropping donor chimerism with cytopenias and/or platelets or red blood cells transfusion requirement).

ELIGIBILITY:
Inclusion Criteria:

1. AML in morphologic remission with intermediate/high-risk features or relapsed disease 1 or 2
2. ALL in morphologic remission with high-risk features or relapsed disease 1 or 2
3. Lymphoid malignancies in CR or PR (e.g. non-Hodgkin's lymphoma, prolymphocytic leukemia, CLL)
4. Myelodysplastic syndromes with <=10% blasts
5. CML in morphologic remission after blast phase or accelerated phase
6. Primary myelofibrosis with <=10% blasts ^morphologic remission is defined as <5% blasts on the bone marrow biopsy. Negative test for donor-specific antibody within 28 days of starting conditioning regimen, or adequate for standard desensitization protocol.

Exclusion Criteria:

1. Non-compliant patients.
2. No appropriate caregivers identified.
3. Uncontrolled medical or psychiatric disorders which may preclude patients to undergo clinical studies (Discretion of the attending physician).
4. Patients with known allergy to DMSO.
5. Pregnant or breastfeeding women

Ages: 4 Weeks to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Severe acute GVHD | 6 years
  Incidence of severe (grade III-IV) acute GVHD <=25% at 100 days
extensive chronic GVHD | 6 years
  Incidence of extensive chronic GVHD <=10% at one year.
donor chimerism | 6 years
  Improvement of donor chimerism by >=15%
Clinical improvement | 6 years
  Clinical improvement, defined as an increase of blood counts with transfusion independence if anemia or thrombocytopenia or freedom for infections if reduced leukocytes

SECONDARY OUTCOMES:
Non-relapse mortality | 6 years
  Rate of one-year non-relapse mortality (NRM).
Disease relapse | 6 years
  Rate of one-year relapse
overall survival | 6 years
  Rate of one-year overall survival (OS).
Absolute neutrophil count | 6 years
  ANC engraftment or increase

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Locatelli F, Lucarelli B, Merli P. Current and future approaches to treat graft failure after allogeneic hematopoietic stem cell transplantation. Expert Opin Pharmacother. 2014 Jan;15(1):23-36. doi: 10.1517/14656566.2014.852537. Epub 2013 Oct 25. PMID 24156789
- [Background] Pasquini MC, Devine S, Mendizabal A, Baden LR, Wingard JR, Lazarus HM, Appelbaum FR, Keever-Taylor CA, Horowitz MM, Carter S, O'Reilly RJ, Soiffer RJ. Comparative outcomes of donor graft CD34+ selection and immune suppressive therapy as graft-versus-host disease prophylaxis for patients with acute myeloid leukemia in complete remission undergoing HLA-matched sibling allogeneic hematopoietic cell transplantation. J Clin Oncol. 2012 Sep 10;30(26):3194-201. doi: 10.1200/JCO.2012.41.7071. Epub 2012 Aug 6. PMID 22869882
- [Background] Roldan E, Perales MA, Barba P. Allogeneic Stem Cell Transplantation with CD34+ Cell Selection. Clin Hematol Int. 2019 Sep 1;1(3):154-160. doi: 10.2991/chi.d.190613.001. eCollection 2019 Sep. PMID 34595425
- [Background] Spohn G, Wiercinska E, Karpova D, Bunos M, Hummer C, Wingenfeld E, Sorg N, Poppe C, Huppert V, Stuth J, Reck K, Essl M, Seifried E, Bonig H. Automated CD34+ cell isolation of peripheral blood stem cell apheresis product. Cytotherapy. 2015 Oct;17(10):1465-71. doi: 10.1016/j.jcyt.2015.04.005. Epub 2015 May 14. PMID 25981397
- Available data/document: Prodigy technical sheet — https://www.miltenyibiotec.com/US-en/products/clinimacs-prodigy.html